CLINICAL TRIAL: NCT05775445
Title: Extremes of Coronary Artery Disease and Normality: Understanding Novel Causative and Protective Factors in the Development of Coronary Artery Disease (CAD Extremes)
Brief Title: Extremes of Coronary Artery Disease and Normality:CAD Extremes
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/2366
Record Dates: First submitted 2023-02-10; First posted 2023-03-20 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 2 tubes of EDTA will be collected per subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 (significant CAD, low risk factors): 1. Evidence of significant CAD
     a. Coronary angiogram or CT coronary angiogram with documented stenosis >=50% in left main or >=70% in major epicardial vessel or major branches (LAD, LCX, RCA)
     AND all of the following
  2. Age </= 45 for males and </= 50 for females
  3. Absence of diabetes mellitus
  4. Absence of tobacco use
  5. No prior CVA or PAD
  Interventions: Procedure: Blood draw
- Group 2 (minor CAD, high risk factors): 1. No evidence of significant CAD
     a. Coronary angiogram or CT coronary angiogram with <50% stenosis in major blood vessel/branch
  2. No prior history of clinical CAD, PAD or CVA
     with one of the
  3. Age >65 with
     1. Diabetes mellitus >5years; or
     2. End Stage Renal Failure (ESRF), regardless of duration or
     3. Framingham risk score > 10%
  4. Diabetes >10 years
  5. End Stage Renal Failure (ESRF) > 5 years
  6. Age >80
  Interventions: Procedure: Blood draw
- Group 3 (signifcant CAD, high risk factors): 1. Evidence of significant CAD with one of the following:
  1. age>65
  2. Diabetes mellitus
  3. End Stage Renal Failure (ESRF)
  4. Framingham risk score >10%
  Interventions: Procedure: Blood draw
- Group 4 Control group: 1. No evidence of significant CAD and all of the following:
  1. Age <55 for males, <65 for females
  2. Absence of diabetes mellitus
  3. Absence of CKD
  4. Absence of tobacco use
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — 2 6ml blood tubes will be collected from patient

SUMMARY:
In the field of cardiovascular medicine, there are two differing groups of patients that remain puzzling to clinicians: patients who are not expected to have coronary artery disease (CAD) yet are diagnosed with significant CAD; and those who are have multiple risk factors for CAD but do not have CAD. Bats exhibit unique phenotypes including long lifespans and likely reduced atherosclerosis. Prior work has identified multiple molecular mechanisms of suppressing the activation of inflammasomes, causally linked to atherosclerosis. The investigators hypothesize there are different molecular markers that confer protection or increased risk for CAD, some of which may be similar to bats. Thus, the aim of this study is to identify molecular markers that contribute to or are protective against acute coronary syndrome (ACS) through analyzing the genetics, peripheral blood and atherosclerotic samples from both extreme patient groups using single-cell RNA sequencing and multi-omics approach. In addition, novel anti-atherosclerotic mechanisms and factors from bat studies will be assessed in the human samples. Identification of novel targets that prevent or cause CAD has the potential to aid in the early identification of high-risk patients and development of new therapeutics to combat this growing epidemic. To conduct this study, patients who have undergone a coronary angiogram or a CT coronary angiogram that fall into the both extremes will be recruited and blood samples will be taken for the above analysis. These will be compared to a group of controls (low risk without disease and high risk with disease).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) imposes much mortality and morbidity worldwide. Large population-based studies in Western cohorts (eg. Framingham Heart Study) have formed the foundations of knowledge on the traditional risk factors of cardiovascular disease. Despite this, large gaps in the knowledge of CVD still exist. The clinical conundrum of the extremes of spectrums of CVD continues to baffle clinicians and researchers alike. These include patients without any major cardiovascular risk factors developing acute coronary syndromes (ACS) at a young age. At the other end of the spectrum, there are not uncommonly patients with "full-house" cardiovascular risk factors with minor or no coronary artery disease.

Similar to the phenotype observed in patients with risk factors with little coronary artery disease, the animal bats exhibit unique phenotypes including long lifespans and likely reduced atherosclerosis. A study has shown that the animal bats are able to have plaque-free arteries despite being on a high-fat diet with high plasma cholesterol, which are associated to the development of atherosclerosis. The pathogenesis of atherosclerosis has been linked to inflammasome activation, an intracellular multi-protein complexes that engage in innate immune defenses. An inflammasome typically consists of a sensor that detects pathogens or danger signals, an adaptor, and an effector that initiates pro-inflammatory responses. Aberrations in inflammasomes have been causally linked to numerous diseases, including viral infections, autoimmune, metabolic, and neurodegenerative diseases. However, no effective treatment options have been established thus far. Importantly, multiple molecular mechanisms of suppressing the activation of inflammasomes, causally linked to atherosclerosis, have already been identified in bats. These include dampened sensors and complementary regulation of the effector and downstream cytokine , which could be protective factors of atherosclerosis. These make bats excellent model for anti-atherosclerosis research.

Recent advancements in technology have led to exciting developments in our understanding of the development and prevention of CVD. The use of "big data" and "deep learning", advancements in genomics, metabolomics, proteomics have the possibility of transforming this field. Recent modern prospective population-based studies (eg. The MURDOCK study) aim to reclassify cardiovascular risk using integrated clinical and molecular biosignatures. However, these studies are based primarily in Western populations. Ethnic differences in CVD exist and currently in Asia, there is a dearth of such advanced data. The aim of this study is thus to identify molecular and inflammasome markers that contribute or are protective against ACS using single-cell sequencing and multi-omics approach, and on top of that, using animal models of bats and mice as comparison to humans. Genomic, metabolomics, proteomics, and scRNA-seq may seek to help answer some of this questions and better improve understanding of the development of CVD, potentially developing novel preventive and management strategies.

The specific aims of the project are as follows:

To use advanced genomic, metabolomics, proteomic and single-cell RNA sequencing (scRNA-seq) analysis to understand novel factors influencing the development of coronary artery disease, as well as protection against coronary artery disease

To assess and validate the novel anti-atherosclerotic mechanisms and factors from bat studies in the human samples

To aid in the development of novel preventive and treatment strategies for coronary artery disease.

Study population

The primary focus will be on two patient groups. Group 1 patients will be recruited to study the novel factors influencing the development of coronary artery disease. This will include patients with known significant coronary artery disease but without any significant major cardiovascular risk factors.

Group 2 patients will be recruited to study the novel factors protective against the development of CAD. This will include patients at high risk of developing CAD but no significant CAD

a group of controls will be recruited (Group 3 and Group 4) for comparison (high risk with CAD and low risk with no CAD). Participants from Group 4 may be obtained from existing registries/cohorts.

Patients will be recruited from two sources:

1. Prospective recruitment from the coronary catheterization lab, CT lab, ward or clinic
2. Retrospective review of angiograms from the coronary catheterization lab and CT coronary angiogram

Informed consent will be obtained. If the patient is agreeable to take part, clinical data will be obtained from his medical records. The patient will also be required to fill up a questionnaire on the patient's demographics, lifestyle and medical history etc. Blood will be obtained from the patients for genetic, proteomic, and metabolic screening.

Other data will be collected if available as part of routine care.

1. Demographic and clinical characteristics data
2. Quality-of-life,
3. Basic blood investigations. Basic blood investigations include: FBC, renal panel, HbA1c, fasting glucose, LFT, fasting lipids, hs-CRP, ESR, ANA, anti-dsDNA, RF, anticardiolipin antibodies, homocysteine, protein C, protein S, thyroid function tests, etc
4. Investigations: ECG, CT, Echo, MRI, holter, nuclear imaging, etc
5. Biobanking and WGS
6. Metabolomic panel

Clinical Follow-up data:

1. Mortality data
2. Stroke/MI/heart failure/Revascularization data
3. Coronary angiograms and other investigations as part of clinical follow up

2. Readmissions 3. Quality of life 4. Costs 5. Other clinical outcomes

These will be obtained from medical records or local, hospital or national databases.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

1. Evidence of significant CAD a. Coronary angiogram or CT coronary angiogram with documented stenosis >=50% in left main or >=70% in major epicardial vessel or major branches (LAD, LCX, RCA)

   AND all of the following
2. Age </= 45 for males and </= 50 for females
3. Absence of diabetes mellitus
4. Absence of tobacco use
5. No prior CVA or PAD

Group 2

1. Evidence of significant CAD

   1. Coronary angiogram or CT coronary angiogram with documented stenosis >=50% in left main or >=70% in major epicardial vessel or major branches (LAD, LCX, RCA)

   AND all of the following
2. Age </= 45 for males and </= 50 for females
3. Absence of diabetes mellitus
4. Absence of tobacco use
5. No prior CVA or PAD

Group 3 1. Evidence of significant CAD with one of the following:

1. age>65
2. Diabetes mellitus
3. End Stage Renal Failure (ESRF)
4. Framingham risk score >10%

Group 4

1. No evidence of significant CAD and all of the following

1. Age <55 for males, <65 for females
2. Absence of diabetes mellitus
3. Absence of CKD
4. Absence of tobacco use

Exclusion Criteria:

1. Prior history of cancer (excludes pre-cancerous lesions)
2. Expected life expectancy less than 1 year
3. Known autoimmune disease
4. Psychiatric illness
5. Chronic lung disease requiring long term medications or oxygen
6. Chronic infective disease, including tuberculosis, hepatitis B and C; and HIV
7. Inability to comply with study protocol
8. Any other acute or chronic medical or physical condition deemed by the investigator to affect study outcomes

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary Artery Disease patients with high risk factors/ low risk factors No Coronary Artery disease but with high risk factors
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Using sequencing analysis to develop treatment to protect against Coronary artery disease | 5 years
  To use advanced genomic, metabolomics, proteomic and single-cell RNA sequencing (scRNA-seq) analysis to understand novel factors influencing the development of coronary artery disease, as well as protection against coronary artery disease
Develop treatment for Coronary artery disease | 5 years
  To aid in the development of novel preventive and treatment strategies for coronary artery disease

CONTACTS AND LOCATIONS:
Overall Officials: Khyung Keong Yeo, Principal Investigator — National Heart Centre
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Participants will be assigned a research ID that only research coordinator and team knows

REFERENCES:
- [Background] Paulin N, Viola JR, Maas SL, de Jong R, Fernandes-Alnemri T, Weber C, Drechsler M, Doring Y, Soehnlein O. Double-Strand DNA Sensing Aim2 Inflammasome Regulates Atherosclerotic Plaque Vulnerability. Circulation. 2018 Jul 17;138(3):321-323. doi: 10.1161/CIRCULATIONAHA.117.033098. No abstract available. PMID 30012706
- [Background] Widmaier EP, Gornstein ER, Hennessey JL, Bloss JM, Greenberg JA, Kunz TH. High plasma cholesterol, but low triglycerides and plaque-free arteries, in Mexican free-tailed bats. Am J Physiol. 1996 Nov;271(5 Pt 2):R1101-6. doi: 10.1152/ajpregu.1996.271.5.R1101. PMID 8945941
- [Background] Alwan A, Maclean DR, Riley LM, d'Espaignet ET, Mathers CD, Stevens GA, Bettcher D. Monitoring and surveillance of chronic non-communicable diseases: progress and capacity in high-burden countries. Lancet. 2010 Nov 27;376(9755):1861-8. doi: 10.1016/S0140-6736(10)61853-3. Epub 2010 Nov 10. PMID 21074258
- [Background] Duewell P, Kono H, Rayner KJ, Sirois CM, Vladimer G, Bauernfeind FG, Abela GS, Franchi L, Nunez G, Schnurr M, Espevik T, Lien E, Fitzgerald KA, Rock KL, Moore KJ, Wright SD, Hornung V, Latz E. NLRP3 inflammasomes are required for atherogenesis and activated by cholesterol crystals. Nature. 2010 Apr 29;464(7293):1357-61. doi: 10.1038/nature08938. PMID 20428172